CLINICAL TRIAL: NCT03526926
Title: A Post-Marketing Observational Study of VYXEOS™ to Assess the Incidence of Infusion-Related Reactions in Adult Patients
Brief Title: A Post-Marketing Observational Study of VYXEOS™
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: CPX351-402
Record Dates: First submitted 2018-05-04; First posted 2018-05-16 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Acute Myeloid Leukemia With Myelodysplasia-Related Changes; Therapy-Related Acute Myeloid Leukemia
Keywords: newly-diagnosed t-AML or AML-MRC
MeSH Terms: interventions — CPX-351

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Vyxeos: A minimum of 50 patients who receive at least one infusion of prescribed VYXEOS.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — VYXEOS is administered as an intravenous (IV) infusion over approximately 90 minutes.
  Other Names: Vyxeos

SUMMARY:
The purpose of this observational study is to provide data on the incidence and severity of infusion-related reactions during and immediately following each infusion of VYXEOS during the first induction.

ELIGIBILITY:
Inclusion Criteria:

1. The decision to prescribe VYXEOS must have been made prior to enrollment in this study and based upon approved US indications and dosing: 44mg/m2 daunorubicin and cytarabine 100 mg/2 on Days 1, 3, and 5.
2. Ability to understand and voluntarily give informed consent and understand the requirements of the registry.
3. Age ≥ 18 years.
4. Initiating VYXEOS therapy for the first time according to the current prescribing information.
5. Initiating VYXEOS therapy for the first time according to standard institutional practice.

Exclusion Criteria:

1. Prior treatment with VYXEOS.
2. Patients receiving any investigational agent other than VYXEOS (e.g., any drug or biologic agent or medical device that has not received approval in the US) or receiving VYXEOS for any indication not currently approved in the US.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A minimum of 50 patients who have received at least one infusion of prescribed VYXEOS at a dose of 44 mg/m2 daunorubicin and 100 mg/m2 cytarabine are planned for this study.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Infusion-Related Reactions on Day 1 | Day 1
  The investigator will assess each AE and indicate if it as an infusion-related reaction.

SECONDARY OUTCOMES:
Incidence of Infusion-Related Reactions Occurring until One Day after the Last Infusion | 1 day after the last infusion
  The number and percentage of patients assessed by the investigator to have had any AEs assessed to be an infusion-related reaction occurring until 1 day after the last infusion.
Changes in Vital Signs | Up to 180 minutes after the start of infusion
  Descriptive statistics for observed vital signs will be provided for each infusion
Incidence of Treatment-emergent Adverse Events (TEAEs) | 1 day after the last infusion
  Treatment-emergent adverse events (TEAEs) are defined as any AE starting after the initiation of the first infusion of VYXEOS

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Franciscan Physician Network Oncology and Hematology Specialists, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina